CLINICAL TRIAL: NCT01233219
Title: Association Between Clinical Effect of Continuous Morphine Administration in Patients After Major Surgery and Pharmacogenetics: Perspective Observational Clinical Study
Brief Title: Association Between Clinical Effect of Continuous Morphine Administration After Surgery and Pharmacogenetics
Status: Withdrawn | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: PT-SM-08-MorfinaContinua-Gene
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia; Surgery
Keywords: systemic morphine analgesia; pharmacogenetics; pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — genes OPRM1, COMT, UGTs, ESR1
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: Homozygous patients for the more frequent allele of the polymorphism A118G of OPRM1 gene
  Interventions: Drug: morphine chlorhydrate
- Group B: Both homozygous and heterozygous patients for the less frequent allele of the polymorphism A118G of OPRM1 gene
  Interventions: Drug: morphine chlorhydrate

INTERVENTIONS:
Drug: morphine chlorhydrate — The drug will be administrated by a bolus 45 minutes before the end of the surgery, with the following modalities: bolus with morphine chlorhydrate 0.15 mg/kg ± 20%. Also acetaminophene 1g and ketoprofen 160 mg (ketorolac 30mg) will be administrated during the operation.
  At the exit of the operative compartment patients will have an continuous infusion for 48h with morphine chlorhydrate 0,02 mg/kg/h.
  Moreover, a rescue dose therapy will be prescribed with ketoprofen 160 mg or ketorolac 30mg (in case of allergy acetaminophene 1g) if NRS<4 maximum x 3 daily.
  Postoperative analgesic treatment is lasting 48h for each patient (between starting of the infusion (T0) and the following 48h).
  Other Names: morfina cloridrato

SUMMARY:
Identification of the genetic polymorphisms that could be correlated either with a better clinical response or with a major predisposition of patients to develop tolerance and/or side effects to the treatment with morphine.

DETAILED DESCRIPTION:
Valuation of the rescue doses necessary to maintain NRS<4 in the first 24 hours post-surgery in the two groups of patients, A e B. Group A: homozygous patients for the more frequent allele of the polymorphism A118G of OPRM1 gene (about 80%); group B: both homozygous and heterozygous patients for the less frequent allele (about 20%).

ELIGIBILITY:
Inclusion criteria:

* Males and females over 18 years, under 75 years, scheduled for postoperative pain control with continuous morphine administration
* HIV negative
* Classification American Society of Anesthesiologists (ASA) I: without systemic disease
* Classification ASA II or III (mild systemic disease or severe systemic disease that limits the activity without invalidity).
* Undergoing abdominal and urologic major surgery (neither urgent nor emergency surgery)
* Signed informed consent

Exclusion criteria:

* Usual assumption of analgesic opioids
* Cognitive alterations nor mental retardation
* Severe hepatic/renal insufficiency (cholinesterase <3000 mU/ml, total bilirubinaemia <2 mg/dl and creatininaemia <1.2 mg/dl)
* Inpatients in intensive therapy, either with sedation and/or mechanic ventilation.
* Allergies to morphine and derivates

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pazients scheduled for major abdominal or urological surgery with postoperative pain control with continuous morphine administration
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of the rescue doses in the two groups homozygous patients for the more frequent allele of the polymorphism A118G of OPRM1 gene; group B: both homozygous and heterozygous patients for the less frequent allele | first 24 h after surgery
  Valuation of the rescue doses necessary to maintain NRS<4 in the first 24 hours post-surgery in the two groups of patients, A e B. Group A: homozygous patients for the more frequent allele of the polymorphism A118G of OPRM1 gene (about 80%); group B: both homozygous and heterozygous patients for the less frequent allele (about 20%).

SECONDARY OUTCOMES:
Variants at the loci OPRM1, COMT, UGTs, ESR1,towards median pain measure | during 24 h postsurgery
  Frequency of the variants at the loci OPRM1, COMT, UGTs, ESR1, both in patients with NRS ≤4 and in those having NRS >4 at least once during 24 hours.
Variants at the loci OPRM1, COMT, UGTs, ESR1,towards median pain measure | period between 24 - 48 h postsurgery
  Frequency of the variants at the loci OPRM1, COMT, UGTs, ESR1, both in patients with NRS ≤4 and in those having NRS >4 at least once during the period between 24-48 hours postsurgery.
Pharmacokinetics of morphine during continuous administration after surgery | 48 h after surgery
  Pharmacokinetic study of both morphine and its principal active and/or toxic metabolites (M3G and M6G).
Detection of the possible side effects. | 72 h postopratively
  Detection of the possible side effects after continuous morphine administration
Detection of the association between M3G/M6G ratio and polymorphisms of UGTs | within 72 h postoperatively
  Detection of the association between M3G/M6G ratio and polymorphisms of UGTs and its possible side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Allegri, MD, Principal Investigator — IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy